CLINICAL TRIAL: NCT00437359
Title: Antiestrogen vs Aromatase Inhibitor After Chemotherapy for Adjuvant Setting: Efficacy of Endocrine Therapy After Chemotherapy in Postoperative Adjuvant Therapy for Breast Cancer
Brief Title: Antiestrogen vs Aromatase Inhibitor After Adjuvant Chemotherapy for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Breast Cancer Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JBCRN-06; UMIN000000610
Record Dates: First submitted 2007-02-18; First posted 2007-02-21 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Drug Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Toremifene; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fareston (Other): Toremifene citrate: 40-mg tablets by mouth once daily.
  Interventions: Drug: Toremifene citrate
- Arimidex (Other): Anastrozole: 1-mg tablets by mouth once daily.
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Toremifene citrate — Toremifene citrate: 40-mg tablets by mouth once daily.
  Other Names: Fareston
  Arms: Fareston
Drug: Anastrozole — Anastrozole: 1-mg tablets by mouth once daily.
  Other Names: Arimidex
  Arms: Arimidex

SUMMARY:
To investigate the benefit of postoperative adjuvant therapy using sequential administration of the hormone, toremifene citrate (TOR) or anastrozole (ANA), after chemotherapy in breast cancer.

DETAILED DESCRIPTION:
To investigate the benefit of postoperative adjuvant therapy using sequential administration of the hormone, toremifene citrate (TOR) or anastrozole (ANA), after chemotherapy in breast cancer.

TOR is reported to be as effective, or more effective, than TAM on both DFS and OS for postoperative adjuvant therapy. The incidence rate and severity of its adverse effects are similar to those of TAM as shown in two clinical trials, the Finnish Breast Cancer Group (FBCG) and the International Breast Cancer Study Group (IBCSG). Although no significant difference was observed in these trials, other studies report that TOR produced a lower number of thromboembolism events compared with TAM, a undesirable side effect seen in patients treated with TAM. Additionally, compared with TAM, TOR showed less endometrial hypertrophy which is induced by estrogen.

Endometrial cancer remains one of the significant problems associated with TAM. A TAM metabolite binds to DNA and forms DNA adducts which damage cells. It is reported that TAM has an expanded ability to form DNA adducts compared with TOR in vitro. A recent study compared endometrial cells collected from patients in which TAM or TOR had been administered. The k-ras gene mutation was investigated in these cases, and it showed that TAM held a higher frequency of gene mutation. Although we still need to discuss whether or not k-ras mutation is directly related to the development of endometrial cancer, TAM seems to have a higher risk of inducing cancer compared with TOR.

In the IBCSG14-93 trials, two chemotherapy protocols were studied subsequent to administration of TOR. They were doxorubicin and cyclophosphamide (AC) and cyclophosphamide, methotrexate, and 5-fluorouracil (CMF). These two chemotherapy protocols were administered in the following sequence: AC four times followed by CMF three times after administration of TOR. The findings revealed that in estrogen-receptor (ER) positive cases, DFS equaled 73% in the TOR group, 65% in the TAM group; hormone receptor (HR=0.80 (0.57-1.11); P=0.18). OS was found to total 88% in the TOR group, 84% in the TAM group; HR=0.78 (0.48-1.27); p=0.32). Although there was no significant difference in two groups, the TOR group has showed somewhat improved survival.

Based on the information provided above, we consider TAM and TOR to have similar efficacy with less adverse effects, and this trial will compare the two drugs, TOR and ANA.

ELIGIBILITY:
Inclusion Criteria:

* Written consent obtained for study participation.
* Breast cancer diagnosed histologically with a breast removed or preserved.
* Positive ER or PR testing by immunohistochemistry (IHC), enzyme immunoassay (EIA) and who meet the criteria of each institution.
* HER2 evaluation.
* Patient Status (PS): 0 or 1.
* Fully functional heart, liver, kidneys, and bone marrow.
* More than one year since last menstruation or tested postmenopausal from estradiol (E2) and follicle-stimulating hormone (FSH) levels based on evaluation standard of each institution.
* Expected to live for at least three months (or longer) after study commencement.

Exclusion Criteria:

* Pregnant or breast feeding.
* Bilateral or inflammatory breast cancer.
* Multiple cancers.
* Life-threatening metastases.
* History of serious hypersensitivity.
* Judged ineligible for the study by the study doctor.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2007-05; Primary Completion 2017-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free rate | The observation period is designated as 10 years from the commencement of treatment.

SECONDARY OUTCOMES:
Survival rate | The observation period is designated as 10 years from the commencement of treatment.
Drug adverse events | The observation period is designated as 10 years from the commencement of treatment.
Bone metabolism markers (BAP, NTx) | Pretreatment, and post-treatment at 3, 6, 12, and 24 months.
BMD (DXA method): Lumbar vertebrae, femoral neck | Pretreatment, and post-treatment at 12 months and 24 months.
Laboratory values of lipid metabolism (TC, LDL, HDL, Lp(a), TG) | Pretreatment, and post-treatment at 3, 6, 12, and 24 months.
Compliance | Compliance status will be entered into the database in the data center every time the study doctor prescribes drugs to the patient (1 to 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Satoru Iwase, MD, Principal Investigator — Department of Palliative Medicine, The University of Tokyo Hospital
Locations (7):
- Japan (7):
  - Kyushu Central Hospital, Fukuoka
  - Kansai Medical University Hirakata Hospital, Hirakata
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima University Hospital, Hiroshima
  - Shinyahashiradai Hospital, Matsudo
  - The University of Tokyo Hospital, Tokyo
  - Nagumo Clinic, Tokyo